CLINICAL TRIAL: NCT00727285
Title: CF Leukocyte Genes as Biomarkers for Novel Therapies
Brief Title: Cystic Fibrosis (CF) Leukocyte Genes as Biomarkers for Novel Therapies
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: NICK07A0
Record Dates: First submitted 2008-07-28; First posted 2008-08-01 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Cystic Fibrosis; Pulmonary Exacerbation
Keywords: Cystic Fibrosis; pulmonary exacerbation; gene expression; biomarker; inflammation; CF pulmonary exacerbation
MeSH Terms: conditions — Cystic Fibrosis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: CF patients followed by the Adult CF Program at National Jewish Health meeting criteria for an acute pulmonary exacerbation.

SUMMARY:
Presently, effectiveness of treatments for CF lung disease is judged by improvement in lung function (FEV1). However, in CF patients, FEV1 can range from severely decreased to normal, and improvements may occur slowly. Thus, clinical trials require many patients over prolonged periods to evaluate medications. As the pace of drug development accelerates, it is no longer possible to test all of the promising candidate therapies using conventional study designs. A sensitive technique for assessing lung inflammation has been developed which uses the expression of genes located in circulating blood cells. Mononuclear cells pass repeatedly through the blood vessels of the lung, and are exposed to many of the inflammatory products that are present in the airways. Over the past 4 years the investigators have identified a small group of candidate genes that are unregulated or downregulated in response to antibiotic treatment. The investigators now propose to prospectively test this method of quantifying lung inflammation in a large group of CF patients undergoing treatment of pulmonary exacerbations. Blood will be sampled before and after antibiotic treatment for a pulmonary exacerbation, and the relative change in gene expression will be compared to improvement in FEV1 and other clinical responses, to determine the utility of this method for use in studies. If successful, this technique could allow for a rapid and noninvasive method to gauge immediate effects by new treatments, and assist caregivers in determining optimal treatment strategies for the individual.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of CF.
2. Age 18 years old or greater.
3. Presentation at the start of treatment for a pulmonary exacerbation of CF.
4. Ability to perform reproducible Pulmonary Function Tests.
5. Willingness to comply with study procedure and willingness to provide written consent.

Exclusion Criteria:

1. Participation in an investigational drug study within one month of enrollment.
2. Presence of a condition or abnormality that, in the opinion of the Principal Investigator (PI), would compromise the safety of the patient or the quality of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CF patients followed by the Adult CF Program at National Jewish Health, who are ≥ 18 years and present with signs and symptoms of an acute pulmonary exacerbation. All subjects will be treated with at least two pathogen specific I.V. antibiotics for a minimum of 10 days, along with standard guidelines for other aspects of care for an acute pulmonary exacerbation. Concomitant use of inhaled antibiotics and systemic steroids will be allowed, and typical co-infections or co-morbidities will not result in exclusion.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The Primary analysis is the change in expression of individual and combinations of mononuclear cell genes, obtained pre- and post-antibiotic therapy. | 14-21 days

SECONDARY OUTCOMES:
Correlation of changes in PBMC gene expression with changes in FEV1 | 14-21 days
Correlation of changes in PBMC gene expression with changes in WBC counts. | 14-21 days

CONTACTS AND LOCATIONS:
Overall Officials: Jerry A Nick, M.D., Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Result] Nick JA, Sanders LA, Ickes B, Briones NJ, Caceres SM, Malcolm KC, Brayshaw SJ, Chacon CS, Barboa CM, Jones MC, St Clair C, Taylor-Cousar JL, Nichols DP, Sagel SD, Strand M, Saavedra MT. Blood mRNA biomarkers for detection of treatment response in acute pulmonary exacerbations of cystic fibrosis. Thorax. 2013 Oct;68(10):929-37. doi: 10.1136/thoraxjnl-2012-202278. Epub 2013 Jun 19. PMID 23783371